CLINICAL TRIAL: NCT04630704
Title: A Feasibility Study Evaluating A Non-Invasive Tissue Perfusion Monitor Utilising Diffuse Speckle Contrast Analysis
Brief Title: Evaluating A Non-Invasive Tissue Perfusion Monitor
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Pedra Technology, PTE LTD (Industry)
Collaborators: Serena Group (Other)
Responsible Party: Sponsor
Other Study IDs: Pedra-001
Record Dates: First submitted 2020-11-05; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Circulatory; Change
Keywords: Microvascular; Perfusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Non vascular repeatibility: This cohort of patients with palpable pulses will be used to test inter- and intra- observer variability for the Pedra system
  Interventions: Device: Pedra
- Non vascular physiology: This cohort of patients with palpable pulses will assess the ability of Pedra to detect perfusion changes in response to physiologic stimuli.
  Interventions: Device: Pedra
- CLTI physiology: This cohort of patients with CLTI will assess the ability of Pedra to detect perfusion changes in response to physiologic stimuli.
  Interventions: Device: Pedra

INTERVENTIONS:
Device: Pedra — Diffuse speckle contrast analysis perfusion system

SUMMARY:
The Pedra perfusion system will be used to assess changes in perfusion in response to physiological stimuli. It will be compared to other standard diagnostics.

DETAILED DESCRIPTION:
The Pedra perfusion system measures microvascular flow through diffuse speckle contrast analysis. It will be used to assess changes in perfusion in response to a number of physiological stimuli. It will be compared to other standard diagnostics including ankle-brachial index, toe-brachial index and transcutaneous oxygen measurement. Measurements will be undertaken in non-vascular patients as well as those with chronic limb threatening ischaemia.

ELIGIBILITY:
Inclusion Criteria:

CLTI cohort

1. At least 40 years old
2. Each patient will have documented arterial occlusive disease within 6 weeks of enrolment as determined by an ankle-brachial index (ABI) < 0.7 but not greater than 1.2, toe-brachial index (TBI) <0.5, skin perfusion pressure (SPP) less than 30mmHg, OR Transcutaneous oxygen measurement (TCOM) < 40mmHg in diabetics and <30mmHg in non-diabetics.
3. The presence of skin breakdown compatible which with an underlying ischemic element (previous minor amputation for gangrene also included) that the Principle Investigator (PI) deems appropriate for the study.
4. Subject has read, understood and signed approved consent, and is willing to participate and comply with the study procedures and requirements.

Non-vascular group

1. At least 40 years old
2. Each patient will have documented palpable foot pulses
3. 21 patients will be free of lower limb oedema and 6 patients will have moderate oedema present
4. Subject has read, understood and signed approved consent, and is willing to participate and comply with the study procedures and requirements.

Exclusion Criteria:

CLTI Cohort

1. Subject on an investigational drug or therapeutic device within 30 days of the study visit, which in the view of the PI may compromise the study results.
2. Presence of a condition that PI considers will compromise the subject's ability to participate in the study.
3. Age <40 or >90
4. Inability to straight leg raise to 30 degrees or tolerate calf cuff occlusion.
5. Has smoked cigarettes/e-cigarettes on the day of testing.
6. Has taken caffeine drinks on the day of testing
7. In the last 3 hours the subject has exercised beyond normal daily walking.
8. Inability to have TBI measured (e.g. absence of toe)
9. Signs of active infection causing localised inflammation on the plantar or dorsal surfaces of the foot
10. Pathological skin conditions that may impair the ability of the adhesive sensor pads to adhere.

Non-vascular Cohort

1. Subject on an investigational drug or therapeutic device within 30 days of the study visit, which in the view of the PI may compromise the study results.
2. Presence of a condition that PI considers will compromise the subject's ability to participate in the study.
3. Age <40 or >90
4. Inability to straight leg raise to 30 degrees or tolerate calf cuff occlusion.
5. Has smoked cigarettes/e-cigarettes on the day of testing.
6. Has taken caffeine drinks on the day of testing
7. In the last 3 hours the subject has exercised beyond normal daily walking.
8. Inability to have TBI measured (e.g. absence of toe)
9. Signs of active infection causing localised inflammation on the plantar or dorsal surfaces of the foot
10. Pathological skin conditions that may impair the ability of the adhesive sensor pads to adhere.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with palpable pulses and patients with chronic limb threatening ischaemia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-12-07 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
The Blood Perfusion Index (unitless number) delta in response to reduction in arterial inflow pressure | Intra-procedure
  The range of change in the Blood Perfusion Index (unitless) in response to physiologic changes in arterial perfusion, in patients with healthy circulation and those with compromised arterial circulation

SECONDARY OUTCOMES:
Reliability of Blood Perfusion Index measurement will be assessed on repeated measures by determination of the correlation coefficient | intra-procedure
  The reliability of measurement of the Blood Perfusion Index will be measured and compared to standard diagnostics
Repeatability of Blood Perfusion Index measurement will be assessed on repeated measures by determination of the correlation coefficient | intra-procedure
  The repeatability of measurement of the Blood Perfusion Index will be measured and compared to standard diagnostics
Sensitivity of Pedra to detect differences in the Blood Perfusion Index between patient subsets | Intra-procedure
  Use of a ROC curve to assess the ability of the Blood Perfusion Index to differentiate between those with healthy circulation and those with arterial disease

IPD SHARING:
Plan to Share IPD: No
No plan to share data